CLINICAL TRIAL: NCT01945515
Title: Robotic-assisted Gait Training Combined With Transcranial Direct Current Stimulation to Maximize Gait Recovery After Stroke: A Double-blind, Randomized, Controlled Trial
Brief Title: Robotic-assisted Gait Training Combined With Transcranial Direct Current Stimulation to Maximize Gait Recovery After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Byung-Mo Oh, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Robot-tDCS-2013
Record Dates: First submitted 2013-09-15; First posted 2013-09-18 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Stroke
Keywords: Stroke; transcranial direct current stimulation; robotic rehabilitation; gait
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Robot + anodal tDCS (Experimental): Robotic-assisted gait training for 45 min after anodal tDCS on impaired motor cortex for 20 min
  Interventions: Device: tDCS; Device: Robotic-assisted gait training
- Robot + sham tDCS (Sham Comparator): Robotic-assisted gait training for 45 min after sham tDCS on impaired motor cortex for 20 min
  Interventions: Device: tDCS; Device: Robotic-assisted gait training

INTERVENTIONS:
Device: tDCS — tDCS will be applied on the primary motor cortex of the lower limb in the impared hemisphere before robotic-assisted gait training. Anodal tDCS will be applied with an intensity of 2mA for 20 min. Sham tDCS will be applied with an intensity of 2mA just for 1 min, after which the current will be slowly tapered down to 0 over a several seconds.
  Other Names: DC-Stimulator Plus (NeuroConn GmbH, Ilmenaus, Germany)
Device: Robotic-assisted gait training — Robotic-assisted gait training with an exoskeletal type robot which simulates normal walking on a treadmill for patients with gait impairments
  Other Names: Walkbot_S (P&S Mechanics Co. Ltd., Seoul, Korea)

SUMMARY:
1. Study objective To evaluate the effect of robotic-assisted gait training combined with transcranial direct current stimulation (tDCS) as compared to that of robotic-assisted gait training on gait function of chronic stroke patients
2. Subjects chronic stroke patients with gait impairment
3. Methods

   * Group 1: Robotic-assisted gait training with anodal tDCS (45 min)
   * Group 2: Robotic-assisted gait training with sham tDCS (45 min)
   * Duration of treatment: 2 weeks, 5 times a week
   * Evaluation: Baseline, 1 day after the treatment, 4 weeks after the treatment

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients who diagnosed by computed tomography or magnetic resonance imaging
* Hemiplegic patients due to unilateral lesion
* Patients in chronic stage after 6 months from stroke onset
* Patients with gait impairment (FAC <= 4)
* Adult (Age >= 18)

Exclusion Criteria:

* Unstable vital sign
* History of seizure or cranial operation
* unable to walk before stroke
* bilateral hemispheric lesions
* metalic implant (cardiac pacemaker, artificial cochlear, etc.)
* severe cognitive deficit, MMSE < 10
* severe aphasic patient who cannot communicate at all

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Functional Ambulatory Category (FAC) | Baseline
  Assesses functional ambulation in patients undergoing physical therapy
Functional Ambulatory Category (FAC) | 1 day after treatment
  Assesses functional ambulation in patients undergoing physical therapy
Functional Ambulatory Category (FAC) | 4 weeks after treatment
  Assesses functional ambulation in patients undergoing physical therapy

SECONDARY OUTCOMES:
10-meter walk test | Baseline
  Time for walking 10 meters
10-meter walk test | 1 day after treatment
  Time for walking 10 meters
10-meter walk test | 4 weeks after treatment
  Time for walking 10 meters
6-min walk test | Baseline
  Walking distance for 6 min
6-min walk test | 1 day after treatment
  Walking distance for 6 min
6-min walk test | 4 weeks after treatment
  Walking distance for 6 min
Modified Rankin's Scale | Baseline
Modified Rankin's Scale | 1 day after treatment
Modified Rankin's Scale | 4 weeks after treatment
Fugl-Meyer assessment scale for lower extremity | Baseline
  Assess the function of lower extremity in stroke patients
Fugl-Meyer assessment scale for lower extremity | 1 day after treatment
  Assess the function of lower extremity in stroke patients
Fugl-Meyer assessment scale for lower extremity | 4 weeks after treatment
  Assess the function of lower extremity in stroke patients
Motor evoked potential | Baseline
  Assess motor pathway from brain cortex to the muscle by transcranial magnetic stimulation
Motor evoked potential | 1 day after treatment
  Assess motor pathway from brain cortex to the muscle by transcranial magnetic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Mo Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea